CLINICAL TRIAL: NCT04094233
Title: Acute Effects of Beet Extract on Autonomic and Cardiovascular Recovery After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Principal Investigator, University of Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UPernambuco14-09
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases; Prevention
Keywords: Beetroot; Heart rate variability; Blood pressure; Strenght Exercise
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beetroot Extract (Experimental): Capsule containing 600mg of beetroot extract.
  Interventions: Dietary Supplement: Beetroot extract; Other: Placebo
- Placebo (Experimental): Capsule containing 600mg of starch.
  Interventions: Dietary Supplement: Beetroot extract; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot extract — Ingestion of 600mg beetroot extract two hours before strength exercise (75% 1RM).
Other: Placebo — Ingestion of 600mg starch two hours before strength exercise (75% 1RM).

SUMMARY:
Dietary NO3 is found in high concentrations in green leafy vegetables and beets. Studies weighing the action of NO3 for ergogenic purposes have found metabolic improvement in skeletal muscle during exercise in hypoxia, lowering blood pressure and increased workload at anaerobic threshold. In a way, the use of nitrate in combination with exercise may assist in autonomic adaptation to multiple stimuli, such as rest, during exercise and during the recovery period. HRV is one of the most practical methods for analyzing the physiological functioning of the ANS, both in the pathological condition of the individual and in the induction of other variables. peak-R (RRI) of consecutive heart beats. This study aims to evaluate the effect of beet extract supplementation in combination with submaximal strength exercise on heart rate variability and cardiovascular parameters of physically active individuals. It is a double-blind randomized crossover clinical trial.

DETAILED DESCRIPTION:
An anamnesis of the participants will be made before the research. Essential information such as name, gender, age, height, BMI will be collected. Anthropometric measurements will be acquired according to the recommendations. Volunteers will be properly informed about the procedures and objectives of this study.

From a pre-established randomization, on the first day of collection volunteers will be allocated to group I (Placebo) or group II (Beet Extract). In the first intervention the volunteers allocated in group I will take a capsule containing 600mg of starch, at the end of this will be provided another capsule containing 600mg of beet extract for the second intervention. Conversely, group II volunteers will ingest a capsule containing 600mg of beet extract in the first intervention, and at the end of the experiment, another capsule containing 600mg of starch will be provided.

Research participants will be advised to consume the capsules within 2 hours of the procedure, adequate time for digestion, absorption and effect on the body. Prior to testing will be asked about the use of caffeine or any other type of substance that is described in the study inclusion and exclusion criteria. Then the collection will proceed.

Participants' blood pressure will be measured before (Rest) and after submaximal strength exercise during the first recovery time (REC1- 00-05 minutes) at 5 1-minute intervals using an aneroid sphygmomanometer (Premium®). and stethoscope (Rappaport®). Korotkoff's first and fifth phase readings were adopted as systolic and diastolic blood pressure, respectively.

Resistance exercise will be performed by performing movements that recruit lower limbs, emphasizing the quadriceps, posterior leg and buttocks. Training intensity will be defined by a subjective test of 1 repetition maximum (1RM). The evaluation will take place at a time before (at least 72 hours) to the data collection, aiming to pre-define and standardize the load that will be used on the day of the experiment. In this sense, the individuals will be oriented to test the load in the 4 proposed physical exercises in a total of 10 maximum repetitions, obtaining 75% of 1 maximum repetition (75% 1RM).

Leg Press 45º - 4 sets x 10 repetitions (75% 1RM) Extender Chair - 4 sets x 10 reps (75% 1RM) Abductor Chair - 4 sets x 10 repetitions (75% 1RM) Guided Squat - 4 sets x 10 repetitions (75% 1RM

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) within the range of Eutrophy (18.5 to 24.9kg / m²)
* Experience with resistance training, uninterrupted for at least 3 months and weekly frequency of 3 sessions or more
* Do not use any medication that may interfere with cardiac autonomic modulation
* Do have no skeletal muscle damage.

Exclusion Criteria:

* Smoking patients
* As well as individuals who have already used anabolic steroids
* Cardiorespiratory diseases
* Neurological disorders
* Other known compromises that prevent the subject from performing the procedures.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Beetroot extract effects on heart rate variability (based on frequency and time domain) | up to 1 year
Blood pressure (mmHg) | up to 1 year
  Beetroot extract effects blood pressure recovery following strength exercise
Heart rate (beats per minute) | up to 1 year
  Beetroot effects heart rate recovery following strength exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Cicero Jonas R Benjamim, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided